CLINICAL TRIAL: NCT06215144
Title: A Phase 2/3 Randomized Double-Blind Placebo Controlled Clinical Trial to Evaluate the Safety and Efficacy of NRCT-101SR in Pediatric Subjects With Attention-Deficit/Hyperactivity Disorder
Brief Title: Study to Evaluate NRCT-101SR in Pediatric Subjects With ADHD
Acronym: ADHD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Neurocentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC-021B
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-03

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Double Blind placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Up to 2,250 mg/day
  Interventions: Drug: NRCT-101SR
- Control Arm (Placebo Comparator): Matching placebo
  Interventions: Drug: NRCT-101SR

INTERVENTIONS:
Drug: NRCT-101SR — NRCT-101SR is a sustained release formulation.
  Other Names: Matching Placebo

SUMMARY:
To evaluate the efficacy and safety of NRCT-101SR compared to placebo in subjects 13-17 years of age with ADHD

DETAILED DESCRIPTION:
a multi-center, randomized, double-blind, placebo-controlled, parallel-arm design, laboratory classroom (LC) clinical trial to evaluate the safety and efficacy of NRCT-101SR (up to to 2,000 mg/day based on LBM) over a 12-week period in approximately 160 pediatric subjects (13-17 years of age) with ADHD.

Selected sites will collect blood samples for PK from a subset of subjects.

The primary endpoint of the study is ADHD Rating Scale (ADHD-RS). The primary analysis will be on effects of 12-week treatment of NRCT-101SR versus placebo on ADHD-RS in subjects with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 13-17 years of age at screening.
2. Has a primary diagnosis of ADHD according to the DSM-5 classification, confirmed with MINI using DSM-5 probes.
3. ADHD-related symptoms - ADHD-RS-5 ≥ 28 in screening and baseline.

   * Baseline score must not change by more than 25% from screening to baseline, except subjects who stop taking ADHD medication after screening may have an increase of more than 25%.
4. Has a minimum score of 5 on the CGI-S at baseline.

Exclusion Criteria:

1. Subject is functioning below an age-appropriate level intellectually, as judged by the Investigator.
2. Lifetime history of severe psychiatric symptoms of major depression requiring hospitalization, bipolar disorder, schizophrenia or schizoaffective disorder, hallucinations, or delusions. Severe comorbid disorders such as PTSD, severe obsessive-compulsive disorder, or other symptomatic presentation that, in the opinion of the examining physician, will contraindicate NRCT-101SR treatment or confound efficacy or safety assessments. Subjects with mild to moderate forms of social phobia or dysthymia, for instance, may be included.
3. History of seizures (other than infantile febrile seizures), any tic disorder (except transient tic disorder and subject has no episodes for at least 1 year), or a current diagnosis of Tourette's Disorder.
4. Recent history (within the past 1 year) of suspected substance abuse or dependence disorder in accordance with DSM-5 criteria.
5. Current abnormal thyroid function as defined as abnormal screening thyroid stimulating hormone. Treatment for at least 3 months with a stable dose of thyroid medication is permitted.
6. History of poor kidney function; corrected estimated glomerular filtration rate (eGFR) < 90 mL/min/m2
7. History of significant gastrointestinal disorders, such as chronic diarrhea, irritable bowel syndrome, ulcerative colitis, Crohn's disease, etc.
8. Female subjects who are pregnant and/or lactating and/or sexually active women of childbearing potential (WOCBP) not agreeing to use birth control methods outlined in inclusion criterion.
9. *A woman is considered fertile following menarche unless permanently sterile; a premenarchal female is not considered a WOBCP).
10. A "yes" answer to "suicidal ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at screening (in the past 12 months).
11. Has history of severe drug allergy or hypersensitivity to the study medication or its excipients.
12. Hypermagnesemia; serum magnesium > 2.5 mg/dL.
13. Hepatic impairment as defined by serum AST, ALT and/or ALP > 1.25 ULN, and/or serum bilirubin > 1.5 ULN.
14. Known history of hepatitis B and/or C.:
15. Is currently participating in another clinical trial or has participated in a clinical trial within 30 days or 5 half-lives of the investigational drug, whichever is longer, prior to the Screening Visit.
16. Currently living in an institutional facility.
17. Severe physical disability not associated with cognitive function that limits ability to complete testing.
18. Known history of symptomatic cardiac disease, advanced atherosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary heart disease, transient ischemic attack or stroke or other serious cardiac problems.
19. Known family history of sudden cardiac death or ventricular arrhythmia.
20. Serious or unstable clinically important systemic illness or disease that, in the judgment of the Investigator, is likely to affect the study assessments, deteriorate, or affect the subject's safety or ability to complete the study, including hepatic (e.g., Child-Pugh grade C), renal, gastroenterological, respiratory, cardiovascular, endocrinologic, immunologic, infectious, or hematologic disorders.
21. Has previously participated in a NRCT-101SR / L-TAMS investigational study.
22. Investigators and their immediate family members are not permitted to participate in the study.
23. Changes in medications or doses of medication as follows:
24. All allowed concomitant medications, supplements, or other substances must be at stable doses for at least 30 days prior to screening and must be kept as stable as medically possible during the trial. For allowed concomitant medications, any dosing change within 30 days of Screening may be allowed if, in the opinion of the Investigator, it will not affect or influence study results.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Core Symptoms/ADHD Rating Scale (ADHD-RS-5) | over 12 weeks
  The ADHD-RS-5 consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with a total score ranging from 0 to 54. Each item has multiple prompts; the highest score that is generated from each prompt should be used as the score for that item. Evaluations will be based on symptoms over the week prior to the administration.

CONTACTS AND LOCATIONS:
Overall Officials: Guosong Liu, MD, PhD, Study Director — Neurocentria, Inc.
Locations (13):
- United States (13):
  - Advanced Research Center, Inc, Anaheim, California
  - Accel Research Sites - Lakeland Clinical Research Unit, Lakeland, Florida
  - Accel Research Sites Network - Maitland, Maitland, Florida
  - Bio-Medical Research LLC, Miami, Florida
  - CenExel ACMR Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - CenExel iRS - iResearch Savannah, Savannah, Georgia
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - Boston Clinical Trials Llc, Boston, Massachusetts
  - Vector Clinical Trials, Las Vegas, Nevada
  - Coastal Carolina Research Center - North Charleston, North Charleston, South Carolina
  - Epic Medical Research - DeSoto, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: No